CLINICAL TRIAL: NCT01202071
Title: A Clinical Pharmacological Study of Rabeprazole Sodium in Japanese Healthy Adult Male Volunteers
Brief Title: A Clinical Pharmacological Study of Rabeprazole Sodium in Japanese Healthy Adult Male Volunteers (Study E3810)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E3810-J081-040
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Rabeprazole; proton pump inhibitor; pharmacokinetics; pharmacodynamics; healthy adult male Japanese subjects
MeSH Terms: interventions — Rabeprazole

ARMS (4):
- Rabeprazole sodium Tablets, 5 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium, 5 mg Tablets
- Rabeprazole sodium Tablets, 10 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium, 10 mg Tablets
- Rabeprazole sodium Tablets, 20 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium, 20 mg Tablets
- Rabeprazole sodium Tablets, 40 mg (two 20 mg Tablets) (Experimental)
  Interventions: Drug: Rabeprazole sodium, 40 mg Tablets (two 20 mg Tablets)

INTERVENTIONS:
Drug: Rabeprazole sodium, 5 mg Tablets — Rabeprazole sodium Tablets, 5 mg administered for 5 days.
  Day 1 and Day 5: participants received a single dose with 200 mL of water in the morning while fasting for 10 hours or longer.
  Day 2 to Day 4: participants received a single dose with 200 mL of water >= 2 hours after the completion of breakfast.
  Other Names: E3810, E3810-J081-040
  Arms: Rabeprazole sodium Tablets, 5 mg
Drug: Rabeprazole sodium, 10 mg Tablets — Rabeprazole sodium Tablets, 10 mg administered for 5 days.
  Day 1 and Day 5: participants received a single dose with 200 mL of water in the morning while fasting for 10 hours or longer.
  Day 2 to Day 4: participants received a single dose with 200 mL of water >= 2 hours after the completion of breakfast.
  Other Names: E3810, E3810-J081-040
  Arms: Rabeprazole sodium Tablets, 10 mg
Drug: Rabeprazole sodium, 20 mg Tablets — Rabeprazole sodium Tablets, 20 mg administered for 5 days.
  Day 1 and Day 5: participants received a single dose with 200 mL of water in the morning while fasting for 10 hours or longer.
  Day 2 to Day 4: participants received a single dose with 200 mL of water >= 2 hours after the completion of breakfast.
  Other Names: E3810, E3810-J081-040
  Arms: Rabeprazole sodium Tablets, 20 mg
Drug: Rabeprazole sodium, 40 mg Tablets (two 20 mg Tablets) — Rabeprazole sodium Tablets, 40 mg (two 20 mg Tablets) administered for 5 days.
  Day 1 and Day 5: participants received a single dose with 200 mL of water in the morning while fasting for 10 hours or longer.
  Day 2 to Day 4: participants received a single dose with 200 mL of water, >=2 hours after the completion of breakfast.
  Other Names: E3810, E3810-J081-040
  Arms: Rabeprazole sodium Tablets, 40 mg (two 20 mg Tablets)

SUMMARY:
The purpose of this study is to compare the pharmacodynamics/pharmacokinetics of 5 mg, 10 mg, 20 mg and 40 mg of Rabeprazole sodium (E3810) when administered repeatedly once daily for 5 days to healthy adult male Japanese participants. This was a single-center, open-label, randomized, four-treatment, four-way crossover study.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult Japanese male between the age of 20-40
* body mass index between 18.5-25

Exclusion Criteria:

* clinically significant abnormal physical examination, vital signs or electrocardiogram
* use of any prescription medication, antacid, nutritional supplement, vitamin preparation, or herb-containing drug within the previous 4 weeks
* use of any non-prescription medication within the previous 1 week
* history of drug or alcohol abuse

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Munesue, Study Director — Japan/Asia Clinical Research Product Creation Unit, Japan Clinical Development, Japan Clinical Development Section
Locations (1):
- Toshima-ku, Tokyo, Japan

REFERENCES:
- [Derived] Hayato S, Hasegawa S, Hojo S, Okawa H, Abe H, Sugisaki N, Munesue M, Horai Y, Ohnishi A. Dose-response relationships of rabeprazole 5, 10, 20, and 40 mg once daily on suppression of gastric acid secretion through the night in healthy Japanese individuals with different CYP2C19 genotypes. Eur J Clin Pharmacol. 2012 May;68(5):579-88. doi: 10.1007/s00228-011-1164-7. Epub 2011 Nov 23. PMID 22108775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 1 center in Japan during the period of 14-Sep-2010 to 2-Dec-2010.
Groups:
- Group A: Rapeprazole 5 mg, Then 10 mg, Then 20 mg, Then 40 mg: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Period I (9 days total): 5 mg; Period II (8 days total): 10 mg; Period III (8 days total): 20 mg; Period IV (8 days total): 40 mg
  Each Period was separated by a >= 6 day washout period.
  Lastly, a follow-up exam, 7 days after Period IV discharge, up to 14 days allowed after discharge.
- Group B: Rapeprazole 10 mg, Then 20 mg, Then 40 mg, Then 5 mg: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Period I (9 days total): 10 mg; Period II (8 days total): 20 mg; Period III (8 days total): 40 mg; Period IV (8 days total): 5 mg
  Each Period was separated by a >= 6 day washout period.
  Lastly, a follow-up exam, 7 days after Period IV discharge, up to 14 days allowed after discharge.
- Group C: Rapeprazole 20 mg, Then 40 mg, Then 5 mg, Then 10 mg: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Period I (9 days total): 20 mg; Period II (8 days total): 40 mg; Period III (8 days total): 5 mg; Period IV (8 days total): 10 mg
  Each Period was separated by a >= 6 day washout period.
  Lastly, a follow-up exam, 7 days after Period IV discharge, up to 14 days allowed after discharge.
- Group D: Rapeprazole 40 mg, Then 5 mg, Then 10 mg, Then 20 mg: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Period I (9 days total): 40 mg; Period II (8 days total): 5 mg; Period III (8 days total): 10 mg; Period IV (8 days total): 20 mg
  Each Period was separated by a >= 6 day washout period.
  Lastly, a follow-up exam, 7 days after Period IV discharge, up to 14 days allowed after discharge.
Period: Overall Study
Arm/Group | Group A: Rapeprazole 5 mg, Then 10 mg, Then 20 mg, Then 40 mg | Group B: Rapeprazole 10 mg, Then 20 mg, Then 40 mg, Then 5 mg | Group C: Rapeprazole 20 mg, Then 40 mg, Then 5 mg, Then 10 mg | Group D: Rapeprazole 40 mg, Then 5 mg, Then 10 mg, Then 20 mg
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Group A, Group B, Group C, Group D: Includes Group A, Group B, Group C, and Group D. Participants received Rabeprazole sodium Tablets for 5 days in each period.
  Group A Period I: 5 mg, Period II: 10 mg, Period III: 20 mg, Period IV: 40 mg
  Group B Period I: 10 mg, Period II: 20 mg, Period III: 40 mg, Period IV: 5 mg
  Group C Period I: 20 mg, Period II: 40 mg, Period III: 5 mg, Period IV: 10 mg
  Group D Period I: 40 mg, Period II: 5 mg, Period III: 10 mg, Period IV: 20 mg
  Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV, a washout period consisted of 6 days or longer between each period.
Arm/Group | Entire Study Population: Group A, Group B, Group C, Group D
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 27.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Baseline Percentage Duration With An Intragastric pH >= 4 During The Entire 24 Hours on Day 1 [Mean (Standard Deviation); unit: Percentage of Time in a 24 Hour Period] — The 24-hour intragastric pH monitoring was performed before the start of administration in Period I. Data was displayed based on the participant's CYP2C19 genotype: CYP2C19-EM are extensive metabolizers who have normal metabolizing capacity. CYP2C19-PM are poor metabolizers with a metabolizing capacity deficiency or remarkably decreased metabolizing capacity.
  Percentage of Time in a 24 Hour Period
    CYP2C19 Extensive Metabolizers 'EM' | 12.57 (7.55)
    CYP2C19 Poor Metabolizers 'PM' | 9.91 (8.50)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Duration With An Intragastric pH >= 4 During The Entire 24 Hours Of Day 5 Administration
Description: The 24-hour intragastric pH monitoring was performed on Day 5 of administration in each study period (Period I-IV). Data was displayed based on the participant's CYP2C19 genotype: CYP2C19-EM are extensive metabolizers who have normal metabolizing capacity. CYP2C19-PM are poor metabolizers with a metabolizing capacity deficiency or remarkably decreased metabolizing capacity.
Time Frame: Day 5 of administration during Period I-IV
Measure: Mean (Standard Deviation); unit: Percentage of Time in a 24 Hour Period
Groups:
- Rabeprazole Sodium 5 mg Tablet: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Rabeprazole sodium 5 mg was received by:
  Group A in Period I; Group B in Period IV; Group C in Period III; Group D in Period II
- Rabeprazole Sodium 10 mg Tablet: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Rabeprazole sodium 10 mg was received by:
  Group A in Period II; Group B in Period I; Group C in Period IV; Group D in Period III
- Rabeprazole Sodium 20 mg Tablet: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Rabeprazole sodium 20 mg was received by:
  Group A in Period III; Group B in Period II; Group C in Period I; Group D in Period IV
- Rabeprazole Sodium 40 mg Tablet: Participants started with a screening period 4 weeks prior to start of administration, followed by study periods I-IV where participants received 5 days of drug administration in each period.
  Rabeprazole sodium 40 mg was received by:
  Group A in Period IV; Group B in Period III; Group C in Period II; Group D in Period I
Arm/Group | Rabeprazole Sodium 5 mg Tablet | Rabeprazole Sodium 10 mg Tablet | Rabeprazole Sodium 20 mg Tablet | Rabeprazole Sodium 40 mg Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
Percentage of Time in a 24 Hour Period
  CYP2C19 Extensive Metabolizers 'EM' (n=16) | 45.63 (19.17) | 57.81 (12.93) | 61.36 (9.72) | 71.52 (12.20)
  CYP2C19 Poor Metabolizers 'PM' (n=8) | 62.51 (14.79) | 71.83 (14.64) | 75.74 (20.62) | 83.08 (11.13)

2. Secondary Outcome: Pharmacokinetic Parameter: Maximal Drug Concentration (Cmax)
Description: Pharmacokinetic parameter: maximal drug concentration (Cmax) measured in nanograms per milliliter (ng/mL) was calculated on Day 1 and Day 5 of administration during each Period (I-IV).
  Data was displayed based on the participant's CYP2C19 genotype: CYP2C19-EM are extensive metabolizers who have normal metabolizing capacity. CYP2C19-PM are poor metabolizers with a metabolizing capacity deficiency or remarkably decreased metabolizing capacity.
Time Frame: Day 1 and Day 5 of administration during Period I-IV
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Rabeprazole Sodium 5 mg Tablet | Rabeprazole Sodium 10 mg Tablet | Rabeprazole Sodium 20 mg Tablet | Rabeprazole Sodium 40 mg Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL
  Day 1: CYP2C19 Extensive Metabolizers 'EM' (n=16) | 137.7 (55.7) | 253.6 (120.2) | 520.0 (267.7) | 1007.6 (513.1)
  Day 5: CYP2C19 Extensive Metabolizers 'EM' (n=16) | 146.0 (56.4) | 382.8 (82.9) | 654.1 (348.4) | 1018.5 (516.9)
  Day 1: CYP2C19 Poor Metabolizers 'PM' (n=8) | 185.1 (79.0) | 434.7 (98.5) | 891.9 (210.8) | 1574.2 (596.6)
  Day 5: CYP2C19 Poor Metabolizers 'PM' (n=8) | 251.9 (55.1) | 508.5 (63.8) | 821.9 (231.7) | 1986.5 (439.1)

3. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t (AUC[0-t])
Description: Pharmacokinetic parameter: Area under the plasma concentration-time curve from time 0 (administration of the drug) to time t (the last quantifiable concentration time point). AUC measured in nanogram hours per milliliter (ng*h/mL) was calculated on Day 1 and Day 5 of administration during each Period (I-IV).
  Data was displayed based on the participant's CYP2C19 genotype: CYP2C19-EM are extensive metabolizers who have normal metabolizing capacity. CYP2C19-PM are poor metabolizers with a metabolizing capacity deficiency or remarkably decreased metabolizing capacity.
Time Frame: Day 1 and Day 5 of administration during Period I-IV (0, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24 hours post-dose)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Rabeprazole Sodium 5 mg Tablet | Rabeprazole Sodium 10 mg Tablet | Rabeprazole Sodium 20 mg Tablet | Rabeprazole Sodium 40 mg Tablet
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL
  Day 1: CYP2C19 Extensive Metabolizers 'EM' (n=16) | 215.5 (88.4) | 429.7 (209.4) | 866.9 (385.6) | 1807.2 (949.2)
  Day 5: CYP2C19 Extensive Metabolizers 'EM' (n=16) | 235.7 (97.1) | 539.1 (199.6) | 993.7 (476.9) | 1929.6 (884.1)
  Day 1: CYP2C19 Poor Metabolizers 'PM' (n=8) | 455.0 (137.7) | 1029.6 (293.9) | 2112.9 (628.8) | 4002.3 (1216.0)
  Day 5: CYP2C19 Poor Metabolizers 'PM' (n=8) | 584.6 (137.1) | 1230.4 (200.0) | 2330.6 (662.9) | 4627.9 (1296.0)

ADVERSE EVENTS:
Arm/Group | Rabeprazole Sodium 5 mg Tablet | Rabeprazole Sodium 10 mg Tablet | Rabeprazole Sodium 20 mg Tablet | Rabeprazole Sodium 40 mg Tablet
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No